CLINICAL TRIAL: NCT03876431
Title: Investigation the Effectiveness of Exercise Device in the Rehabilitation of Total Knee Arthroplasty
Brief Title: Exercise Device in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Zeynal YASACI, Research Assistant; Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/01/2018-17939
Record Dates: First submitted 2019-02-21; First posted 2019-03-15 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Total Knee Arthroplasty; Total Knee Replacement
Keywords: Knee prosthesis; Physiotherapy; Range of motion
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Exercise Group (Active Comparator): Only traditional exercises will be performed in the early post-op period.
  Interventions: Other: Exercise
- Easy-Flex Group (Experimental): Easy-Flex group will be treated with the Easy-Flex device in addition to the traditional exercise program.
  Interventions: Device: Easy-Flex; Other: Exercise

INTERVENTIONS:
Device: Easy-Flex — The Easy-Flex device will be used to increase knee flexion and extension ROM.
  Arms: Easy-Flex Group
Other: Exercise — After total knee replacement surgery, exercise program including strengthening, stretching and patient training will be applied.

SUMMARY:
Total knee arthroplasty is performed in patients with advanced stages of osteoarthritis who can not respond to conservative treatment, in order to reduce pain, increase range of motion, and improve function and quality of life. Continuous passive motion device continues to be used in many clinics, although it has been shown that there is no effect in total knee arthroplasty rehabilitation. The aim of the study was to assess the clinical effects of the knee exercise device on pain, ROM and function and quality of life in total knee arthroplasty rehabilitation.

DETAILED DESCRIPTION:
Volunteers with total knee arthroplasty according to the criteria of inclusion, who will be operated in Istanbul University Istanbul Medical Faculty Orthopedics and Traumatology Department will be included this study. Participants will be randomly allocated 2 groups: easy-flex group and traditional exercise group. Exercise group will be treated with the traditional exercise program and the Easy-Flex group will be treated with the Easy-Flex device in addition to the traditional exercise program.

ELIGIBILITY:
Inclusion Criteria:

Patients with TKA surgery due to the diagnosis of knee OA Between the ages of 45-80 years Patients with no difference over 5 cm in the extremity before and after surgery

Exclusion Criteria:

Revision TKA, Previous unicompartmental arthroplasty or tibial osteotomy, Hemophilia, Uncontrolled hypertension Rheumatic diseases, Lower extremity fractures and tumors, Neurological diseases leading to muscle weakness in the lower limbs, Patients with emotional and cognitive problems

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change range of motion | Assessment is performed at pre-op and post-op second and sixth weeks rehabilitation program.
  Range of motion of knee flexion and extension

SECONDARY OUTCOMES:
NPRS (Numerical Pain Rating Scale) | Assessment is performed at pre-op and post-op second and sixth weeks rehabilitation program.
  The levels of pain intensity measured using NPRS (Numerical Pain Rating Scale). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
WOMAC | Assessment is performed at pre-op and post-op second and sixth weeks rehabilitation program.
  Measure of symptoms and physical disability
Satisfaction levels of the patients | At sixth week
  Satisfaction levels of the patients with Global Rating of Change Score
Short Form 12 (SF-12) | Assessment is performed at pre-op and post-op second and sixth weeks rehabilitation program.
  SF-12 is used to assess physical and mental health-related quality of life. The high scores are positively correlated with the high quality of life.
10 meter walking test | Assessment is performed at pre-op and post-op second and sixth weeks rehabilitation program.
  To test comfortable or maximal walking speed
5 sit to stand | Assessment is performed at pre-op and post-op second and sixth weeks rehabilitation program.
  To measure performance of lower extremity

CONTACTS AND LOCATIONS:
Overall Officials: Derya Çelik, Professor, Study Director — Istanbul University Faculty of Health Sciences; Zeynal Yasacı, Principal Investigator — Istanbul University Faculty of Health Sciences
Locations (1):
- Istanbul Faculty Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No